CLINICAL TRIAL: NCT02457923
Title: Mobile Health Solutions to Help Community Providers Promote Maternal & Infant Nutrition & Health - A Community-based Cluster RCT in Rural India to Evaluate M-SAKHI for Use by ASHAs to Reduce Malnutrition in Infants up to 24 Months
Brief Title: Mobile -Solutions Aiding Knowledge for Health Improvement
Acronym: M-SAKHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lata Medical Research Foundation, Nagpur (Other)
Collaborators: ADVANCING REDUCTION IN MORTALITY AND MORBIDITY OF MOTHERS, CHILDREN AND NEONATES (Unknown); Dimagi Inc. (Industry); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02_MSAKHI
Record Dates: First submitted 2015-05-14; First posted 2015-05-29 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Under Nutrition
Keywords: mobile phone counselling; infant feeding; nutrition
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone counselling (Experimental): The intervention will include:
  * An "App" for real time data collection of mothers by ASHAs, data transfer, and, display of counselling messages and health video during ASHAs monthly home visit.
  * Weekly voice and text messages from server at a prescribed time to provide targeted information on infant feeding counselling.
  * Server generated reminders and alerts, delivered to the mother, ASHA and ANM.
  * An "App" for field supervisor to monitor ASHAs
  * Women will receive fortnightly mobile phone counselling calls by an ANM at times they recommend. Need based counselling will also be provided
  Interventions: Other: Mobile phone counselling
- Usual health care services (No Intervention): The control clusters to receive usual health care services at PHC. The existing data collection methods will be continued in these clusters. Routine IYCF counseling is provided in existing level of care and its frequency is consistent with the visit schedule described in the intervention group: at antenatal clinics; at delivery; and at immunization clinics postnatal.

INTERVENTIONS:
Other: Mobile phone counselling — i) Data collection and counselling by ASHA using the cell application (App) developed by CommCare Dimagi ii) Mobile phone counselling iii) Routine counselling schedules
  Other Names: Mobile app for data collection
  Arms: Mobile phone counselling

SUMMARY:
Using a community-based, cluster randomized controlled trial design (cRCT) the investigators will examine the impact of an integrated "m-health package -(M- SAKHI) for mothers on appropriate infant feeding practices, starting in the first / second trimester of pregnancy to 24 months after delivery, to improve child feeding practices and child growth, and reduce the prevalence of undernutrition in their children. This will result in two treatment groups. The clusters for the trial will be villages under the administrative area of ASHAs (Accreditated Social Health Activists). Villages with a population of 1000- 2000 (ranging from 751 to 2000) with 1 ASHA will be randomized to receive intervention (intervention villages) or continue existing delivery of care (control villages). The data will be collected using a longitudinal design because the investigators want to study the impact of intervention on the mothers starting at pregnancy until her infant is 24 month old.

DETAILED DESCRIPTION:
a. Study design: Using a community-based, cluster randomized controlled trial design (cRCT) the investigators will examine the impact of an integrated "m-health package - (M- SAKHI) for mothers on appropriate infant feeding practices, starting in the first / second trimester of pregnancy to one year after delivery, to improve child feeding practices and child growth, and reduce the prevalence of undernutrition in their children. This will result in two treatment groups (see diagram). The clusters for the trial will be villages under the administrative area of ASHAs. Villages with a population of 1000- 2000 (ranging from 751 to 2000) with single ASHA will be randomized to receive either this intervention (intervention villages) or continue with existing delivery of care (control villages). Selecting a single village per ASHA criteria will reduce the chances of contamination of study groups. The data will be collected using a longitudinal design because the investigators want to study the impact of intervention on the mothers starting at pregnancy until her infant is 24 month old. This is preferred to a cross sectional design to reduce the impact due to migration of mothers in or out of the clusters, who may not receive the intervention as planned. Cross sectional surveys are better suited if a before and after intervention design is used. Lastly on-going government programs can contaminate the intervention in a before-after cross section design. However in a CRCT, the government programs will be present in both study and control clusters, so the additional impact of the intervention can be evaluated. Additionally, growth velocity and development of an infant whose mother is receiving the intervention can also be evaluated using a longitudinal design.

This design will control for potential confounding factors (Observed and unobserved) because an adequate number of clusters (292 villages) will be randomly allocated to the treatment groups. This random allocation of treatments by villages will reduce selection bias that would arise if better performing PHCs with favorable local conditions were purposely selected. Contamination of intervention will be constrained by the administrative and geographic separation of the villages, and by buffer areas.

The outcome assessments will be made by field research officers (FROs) on a cohort of 2,728 mother-infant dyads (1,364 in each treatment group) measured at baseline and at follow up visits. There will be follow-up assessments every trimester during pregnancy and every month from birth until the children are 12 months of age, and then every three or 6 months till 24 months. Three of these assessments (when infants are 15,18 & 24 months) will be made after the education intervention has ceased in order to assess the sustained impact on the prevalence of child stunting and infant feeding practices (see evaluation plan or details). The investigators expect a likely high correlation between baseline and follow up outcome measures, and low loss to follow up, thus making this approach the most efficient study design.

In this cRCT the interventions will be allocated at a community level, but the outcome assessments will be at the individual level. This is the best comparative design for the proposed interventions, which if delivered to individual mothers would most likely lead to contamination of the intervention in the densely populated rural village communities.

The proposed field area will be the centrally located villages in the catchment areas of Indian Government, PHC in 3 districts (Nagpur, Bhandara and Wardha) of eastern Maharashtra (see Map).There are around 28 PHCs.Each Primary Health Centre (PHC) covers an average population of 30,000 with an average of 30 villages. The administrative area under an ASHA is villages with population of 1000-200 (range of 751 to 2000).

As per the investigators' experience in the Maternal and Neonatal Health (MNH) Registry, the Crude Birth Rate (CBR) of the study area is 16.4 per 1000 population, thus expected or projected number of ante-natal cases (ANC) per thousand populations would be 18 per year considering 10 per cent pregnancy wastage.

At any given point of time, 60 per cent ANCs (11) will be available per thousand population, of which 6 will be up to 20 weeks of gestation. An additional 6 can be registered during next 3 months of enrollment period.

Using standard formulae, the sample size required would be 2,728 mother-infant pairs (1,364 per group) from 292 clusters .This sample would provide 90% power to detect a 15% relative reduction in stunting. Based on prior experience the investigators estimate that after accounting for probable cases of loss to follow-up and delivery outside the study area, about 70 percent of ANCs would be available for inclusion in the study. Thus 8 ANCs per 1000 population would be available for inclusion in the study and a population of 341000 needs to be covered to get required number (2728) subjects.

The unit of randomization will be the ASHA who provides her services to a village with a average population of 1000-2000 (ranging from 751 - 2000) persons. Using a computerized random number generator the investigators will randomize 146 ASHA (1 ASHA per village) to deliver services to pregnant women till her infant is 12 months using the M-SAKHI intervention in addition to the exiting services (intervention group), and, 146 to control group i.e routine provision of services or existing level of service delivery (uniform allocation), across each geographic area. The random allocation sequence will be generated using Stata® software.

All efforts will be made to enroll the women in their first / second trimester (up to 20 weeks of gestation). In both arms, to encourage women to enroll as early as possible, the eligible couples will be identified by ASHA and incentivized by home pregnancy test kits, so that they could report as soon they missed their periods. The average expected number of births for the population covered by 292 villages in the PHCs over 12 months would be 3000, which would be more than required for trial recruitment, thus confirming the feasibility of the sampling scheme.

ELIGIBILITY:
Inclusion Criteria:

* A population of 1000-2000 (ranging from 751-2000) persons and geographically at a distance from other selected villages
* Within 100 kms distance from the study co-ordinating centre
* With good cell phone network connectivity (>70%)
* At least 80% of households with at least one cell phone
* Staff of the public health system willing to participant in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2728 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the percentage of stunted infants | 36 months
  Changes in the percentage of stunted infants (height-for-age <-2 Z) at 6, 12, 15,18 and 24 months as measured in follow up assessments starting from birth

OTHER OUTCOMES:
Mean cost per stunted infant prevented | 36 months
  Cost effectiveness of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Archana B Patel, MD, PhD, Principal Investigator — Lata Medical Research Foundation
Locations (1):
- Public Health system, Nagpur, Maharashtra, India

REFERENCES:
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Institute for Health Metrics and Evaluation. GBD Heatmap. 2013. http://www.healthmetricsandevaluation.org/gbd/visualizations/gbdheatmap (accessed 10th March 2013).
- [Background] Stevens GA, Finucane MM, Paciorek CJ, Flaxman SR, White RA, Donner AJ, Ezzati M; Nutrition Impact Model Study Group (Child Growth). Trends in mild, moderate, and severe stunting and underweight, and progress towards MDG 1 in 141 developing countries: a systematic analysis of population representative data. Lancet. 2012 Sep 1;380(9844):824-34. doi: 10.1016/S0140-6736(12)60647-3. Epub 2012 Jul 5. PMID 22770478
- [Background] Christian P, Lee SE, Donahue Angel M, Adair LS, Arifeen SE, Ashorn P, Barros FC, Fall CH, Fawzi WW, Hao W, Hu G, Humphrey JH, Huybregts L, Joglekar CV, Kariuki SK, Kolsteren P, Krishnaveni GV, Liu E, Martorell R, Osrin D, Persson LA, Ramakrishnan U, Richter L, Roberfroid D, Sania A, Ter Kuile FO, Tielsch J, Victora CG, Yajnik CS, Yan H, Zeng L, Black RE. Risk of childhood undernutrition related to small-for-gestational age and preterm birth in low- and middle-income countries. Int J Epidemiol. 2013 Oct;42(5):1340-55. doi: 10.1093/ije/dyt109. Epub 2013 Aug 6. PMID 23920141
- [Background] Dewey KG, Brown KH. Update on technical issues concerning complementary feeding of young children in developing countries and implications for intervention programs. Food Nutr Bull. 2003 Mar;24(1):5-28. doi: 10.1177/156482650302400102. PMID 12664525
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Patel A, Badhoniya N, Khadse S, Senarath U, Agho KE, Dibley MJ; South Asia Infant Feeding Research Netwoork. Infant and young child feeding indicators and determinants of poor feeding practices in India: secondary data analysis of National Family Health Survey 2005-06. Food Nutr Bull. 2010 Jun;31(2):314-33. doi: 10.1177/156482651003100221. PMID 20707236
- [Background] Patel A, Pusdekar Y, Badhoniya N, Borkar J, Agho KE, Dibley MJ. Determinants of inappropriate complementary feeding practices in young children in India: secondary analysis of National Family Health Survey 2005-2006. Matern Child Nutr. 2012 Jan;8 Suppl 1(Suppl 1):28-44. doi: 10.1111/j.1740-8709.2011.00385.x. PMID 22168517
- [Background] Bhutta ZA, Ahmed T, Black RE, et al. Maternal and Child Undernutrition 3: What works? Interventions for maternal and child undernutrition and survival. Child-Care Health and Development 2008; 34(3): 404-.
- [Background] Shrimpton R, Victora CG, de Onis M, Lima RC, Blossner M, Clugston G. Worldwide timing of growth faltering: implications for nutritional interventions. Pediatrics. 2001 May;107(5):E75. doi: 10.1542/peds.107.5.e75. PMID 11331725
- [Background] Victora CG, de Onis M, Hallal PC, Blossner M, Shrimpton R. Worldwide timing of growth faltering: revisiting implications for interventions. Pediatrics. 2010 Mar;125(3):e473-80. doi: 10.1542/peds.2009-1519. Epub 2010 Feb 15. PMID 20156903
- [Background] Mathers CD, Boerma T, Ma Fat D. Global and regional causes of death. Br Med Bull. 2009;92:7-32. doi: 10.1093/bmb/ldp028. PMID 19776034
- [Background] Jones G, Steketee RW, Black RE, Bhutta ZA, Morris SS; Bellagio Child Survival Study Group. How many child deaths can we prevent this year? Lancet. 2003 Jul 5;362(9377):65-71. doi: 10.1016/S0140-6736(03)13811-1. PMID 12853204
- [Background] International Institute for Population Sciences (IIPS), ORC Macro. National Family Health Survey (NFHS-3), 2005-06: India. Mumbai: IIPS 2006; Vol. 1.
- [Background] International Institute for Population Sciences (IIPS). Comprehensive Nutrition Survey in Maharashtra (CNSM). Fact Sheet. 2012
- [Background] Haider R, Ashworth A, Kabir I, Huttly SR. Effect of community-based peer counsellors on exclusive breastfeeding practices in Dhaka, Bangladesh: a randomised controlled trial [see commments]. Lancet. 2000 Nov 11;356(9242):1643-7. doi: 10.1016/s0140-6736(00)03159-7. PMID 11089824
- [Background] Hayes RJ, Moulton LH. Cluster randomised trials: CRC Press London; 2009
- [Background] World Health Organisation. Ottawa Charter for Health Promotion. 1986. www.who.int/hpr/NPH/docs/ottawa_charter_hp.pdf (accessed 13th March, 2013 2013).
- [Background] Lohman T, Roache A, Martorell R. Anthropometric standardization reference manual. Medicine & Science in Sports & Exercise 1992; 24(8): 952.
- [Background] World Health Organization. Nutrition for Health. WHO child growth standards: growth velocity based on weight, length and head circumference: Methods and development: World Health Organization; 2009.
- [Background] Gopalan C, Sastri BR, Balasubramanian S. Nutritive value of Indian foods. Hyderabad: National Institute of Nutrition 1971
- [Background] Filmer D, Pritchett LH. Estimating wealth effects without expenditure data--or tears: an application to educational enrollments in states of India. Demography. 2001 Feb;38(1):115-32. doi: 10.1353/dem.2001.0003. PMID 11227840
- [Background] Borghi J, Thapa B, Osrin D, Jan S, Morrison J, Tamang S, Shrestha BP, Wade A, Manandhar DS, Costello AM. Economic assessment of a women's group intervention to improve birth outcomes in rural Nepal. Lancet. 2005 Nov 26;366(9500):1882-4. doi: 10.1016/S0140-6736(05)67758-6. PMID 16310555
- [Background] Department of Comupter Science and Engineering, Change. Open Data Kit. 2013. www.opendatakit.org (accessed 15th March 2013).
- [Background] Penny ME, Creed-Kanashiro HM, Robert RC, Narro MR, Caulfield LE, Black RE. Effectiveness of an educational intervention delivered through the health services to improve nutrition in young children: a cluster-randomised controlled trial. Lancet. 2005 May 28-Jun 3;365(9474):1863-72. doi: 10.1016/S0140-6736(05)66426-4. PMID 15924983
- [Background] Murray DM. Design and analysis of group-randomized trials: Oxford University Press, USA; 1998.
- [Background] Briggs A, Sculpher M, Claxton K. Decision modelling for health economic evaluation. OUP Catalogue 2011.